CLINICAL TRIAL: NCT03136627
Title: A Phase 1b/2, Open-Label, Multi-Center Study of Tivozanib in Combination With Nivolumab in Subjects With Metastatic Renal Cell Carcinoma
Brief Title: Phase 1/2 Study of Tivozanib in Combination With Nivolumab in Subjects With RCC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-16-119
Record Dates: First submitted 2017-04-07; First posted 2017-05-02 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Carcinoma, Renal Cell
Keywords: RCC, Tivozanib, Nivolumab, Metastatic Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — tivozanib; Nivolumab

STUDY DESIGN:
Intervention Model Description: Tivozanib in Combination with Nivolumab
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tivozanib (AV-951) plus Nivolumab (Experimental): Tivozanib plus Nivolumab:Tivozanib will be administered once daily for 3 weeks followed by 1 week off. Nivolumab will be administered every 2 weeks starting on Day 1.
  Interventions: Drug: Tivozanib; Drug: Nivolumab

INTERVENTIONS:
Drug: Tivozanib — Tivozanib (AV-951): Phase 1b study and Phase 2a study: Subjects will receive 1 dose of tivozanib daily for 21 days followed by a 7 day rest period (1 cycle = 4 weeks).
  Other Names: AV-951
Drug: Nivolumab — Nivolumab: Phase 1b study and Phase 2a study: All subjects will receive IV nivolumab 240 mg every 2 weeks administered over 1 hour.
  Other Names: Opdivo (anti-PD-1 monoclonal antibody)

SUMMARY:
This study will evaluate the safety, tolerability, dose-limiting toxicities, MTD, and preliminary anti-tumor activity of tivozanib in combination with nivolumab in subjects with metastatic renal cell cancer. This will use a standard '3+3' dose-escalation trial design. A cohort of 3 subjects will be enrolled at each dose level. If 1 of 3 subjects experiences a DLT during Cycle 1, that dose level will be expanded to 6 subjects. If 0 of 3 or ≤ 1 of 6 subjects experience a DLT during Cycle 1, escalation to the next dose will occur. If ≥ 2 of 6 subjects experience a DLT during Cycle 1, dose escalation will stop and the prior dose will be considered the MTD. This is a validated trial design for Phase 1 trials.

Following completion of the dose-escalation cohorts and determination of MTD, an expansion cohort of up to 20 subjects may be enrolled at MTD to further evaluate safety, tolerability, and preliminary anti-tumor activity of tivozanib in combination with nivolumab in the same target population.

DETAILED DESCRIPTION:
Tivozanib hydrochloride (tivozanib; previously known as AV-951 and as KRN951) has the chemical name (N-{2-Chloro-4-[(6,7-dimethoxy-4-quinolyl)oxy]phenyl}-N'-(5-methyl-3-isoxazolyl)urea hydrochloride monohydrate. Tivozanib is a novel and potent vascular endothelial growth factor (VEGF) receptor tyrosine kinase inhibitor (VEGFR TKI) that has demonstrated significant anti-tumor effects in pre clinical experiments [1]. Tivozanib inhibits phosphorylation of VEGF receptors (VEGFR) -1, -2 and -3 at picomolar concentrations (IC50 of 0.21, 0.16 and 0.24 nM respectively), and inhibits c-Kit and platelet derived growth factor receptor (PDGFR) at 10-times higher concentrations (IC50 of 1.63 and 1.72 nM respectively).

Based on its biochemical profile, tivozanib appears to be one of the most potent and selective VEGF tyrosine kinase inhibitor in clinical development. Other agents used for treatment of renal cell carcinoma (RCC) such as sunitinib and sorafenib inhibit multiple tyrosine kinases in addition to the VEGF receptor tyrosine kinase, leading to off-target toxicities such as fatigue, hand-foot syndrome, stomatitis, and neutropenia. The adverse event (AE) profile of tivozanib demonstrates that it is a selective VEGF tyrosine kinase inhibitor, with reduced off-target toxicities.

Nivolumab is a fully human IgG4 programmed death 1 (PD-1) immune checkpoint inhibitor antibody that selectively blocks the interaction between PD-1, which is expressed on activated T cells, and PD-1 ligand 1 (PD-L1) and 2 (PD-L2) which are expressed on immune cells and tumor cells. Interaction between PD-1 and PD-L1 or PD-L2 normally results in the inhibition of the cellular immune response. Nivolumab has shown activity in renal cell carcinoma. [2]

This study is designed to test the hypothesis that tivozanib can be combined with nivolumab for the treatment of patients with renal cell carcinoma. The purpose of the study is to determine the maximum dose of tivozanib that can be safely combined with nivolumab, and to evaluate the safety profile and tolerability of this combination. Given the different mechanisms of action and a lack of overlapping toxicities this combination may provide an alternative therapy to patients with renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18-year-old
2. Histologically or cytologically documented renal cell carcinoma with a clear cell component, except in Phase 1b, where any histology will be permitted
3. Metastatic renal cell carcinoma. Measurable or evaluable disease by RECIST 1.1 criteria
4. No prior exposure to tivozanib or nivolumab
5. ECOG performance status ≤ 1 (see Appendix A) and life expectancy ≥ 3 months.
6. Signed and dated written informed consent
7. Sexually active pre-menopausal female subjects and female partners of male subjects must use adequate contraceptive measures, while on study and for at least 160 days after the last dose of study drug. Sexually active male subjects must use adequate contraceptive measures, while on study and for at least 160 days after the last dose of study drug. All fertile male and female subjects and their partners must agree to use a highly effective method of contraception. Effective birth control includes (a) intrauterine device (IUD) plus one barrier method; or (b) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). Note: Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are not considered effective for this study.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Subjects with symptomatic CNS metastases. Subjects with treated brain metastases that have remained stable for at least 3 months without steroids are allowed. Subjects with signs or symptoms or history of brain metastasis must have a CT or MRI scan of the brain within 1 month prior to the start of protocol therapy. Subjects with spinal cord or nerve root compression who have completed treatment at least 4 weeks before the start of protocol therapy and are stable without steroid treatment for at least one week before start of protocol therapy are allowed. Subjects with leptomeningeal metastases are not allowed.
3. Any of the following hematologic abnormalities:

   * Hemoglobin < 9.0 g/dL
   * ANC < 1500 per mm3
   * Platelet count < 100,000 per mm3
4. Any of the following serum chemistry abnormalities:

   * Total bilirubin > 1.5 × ULN (>2.5 mg/dL in patients with Gilbert's syndrome)
   * AST or ALT > 2.5 × ULN (or > 5 × ULN for subjects with liver metastasis)
   * Alkaline phosphatase > 2.5 × ULN (or > 5 × ULN for subjects with liver or bone metastasis)
   * Serum creatinine > 1.5 × ULN
   * Proteinuria > 2.5 g/24 hours or 3+ with urine dipstick
   * Any other ³ Grade 3 laboratory abnormality at baseline (other than those listed above)
5. Significant cardiovascular disease, including:

   * Clinically symptomatic heart failure. Subjects with a history of heart failure must have an ECHO or MUGA scan to document left ventricular ejection fraction (LVEF) > 45% prior to start of protocol therapy
   * Uncontrolled hypertension: blood pressure >150/95 mmHg on more than 2 antihypertensive medications, on two consecutive measurements obtained at least 24 hours apart. Subjects with a history of hypertension must have been on stable doses of anti-hypertensive drugs for ≥ 2 weeks prior to start of protocol therapy.
   * Myocardial infarction within 3 months prior to start of protocol therapy
6. Subjects with delayed healing of wounds, ulcers, and/or bone fractures
7. Serious/active infection or infection requiring parenteral antibiotics
8. Inadequate recovery from any prior surgical procedure; major surgical procedure within 4 weeks prior to start of protocol therapy.
9. Inability to comply with protocol requirements
10. Subjects with a "currently active" second primary malignancy other than non-melanoma skin cancers. Subjects are not considered to have a "currently active" malignancy if they have completed anti-cancer therapy and have been disease free for > 2 years.
11. Known concomitant genetic or acquired immune suppression disease such as HIV
12. Treatment with systemic hormonal therapy within 3 weeks prior to start of protocol therapy, with the exception of:

    * Hormonal therapy for appetite stimulation or contraception
    * Nasal, ophthalmic, inhaled and topical steroid preparations
    * Oral replacement therapy for adrenal insufficiency
    * Low-dose maintenance steroid therapy (equivalent of prednisone 10mg/day) for other conditions
    * Hormone replacement therapy
13. Herbal preparations/supplements (except for a daily multivitamin/mineral supplement not containing herbal components) or CYP3A4 inhibitors or inducers (see Appendix B) within 2 weeks prior to start of or during protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of tivozanib administered orally in combination with Nivolumab in subjects with advanced renal cell carcinoma. | 28 days (1 Cycle)
  A traditional escalation rule, also known as "3 + 3" rule, will be used for this study. Subjects are treated in groups of 3 with each receiving the same dose. If none of the 3 subjects experience a DLT within Cycle 1, the next group of 3 subjects receives the next higher dose, otherwise, the group will expand to 6 subjects treated at the same dose level. If ≤ 1 of the 6 subjects treated at that dose level experience a DLT within Cycle 1, the trial will continue to the next higher dose level. If ≥ 2 of the 6 experience a DLT at the dose level within Cycle 1, then escalation stops at that level and the prior dose level will be considered the MTD. If MTD is not identified and both dose levels are tolerated, 1.5 mg will be considered the recommended Phase II dose (RP2D) for the expansion.

SECONDARY OUTCOMES:
Disease status will be summarized by cycle and dose group, including changes from baseline. | Every 3 months during the first year [beginning from the date of the last scan performed prior to treatment discontinuation], and every 6 months thereafter (up to 24 months) until disease progression or start of another anti-cancer therapy.
  Upon determination of MTD, up to 20 additional subjects with measurable disease will be enrolled in the MTD Expansion Cohort for an expanded assessment of safety and activity.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Bordeaux Hospital University Center (CHU), Bordeaux
  - Center Léon Bérard, Lyon
  - Centre Paul Strauss, Strasbourg
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Albiges L, Barthelemy P, Gross-Goupil M, Negrier S, Needle MN, Escudier B. TiNivo: safety and efficacy of tivozanib-nivolumab combination therapy in patients with metastatic renal cell carcinoma. Ann Oncol. 2021 Jan;32(1):97-102. doi: 10.1016/j.annonc.2020.09.021. Epub 2020 Sep 30. PMID 33010459